CLINICAL TRIAL: NCT05959447
Title: A Phase 1, 2-part, Open-label, Fixed-sequence Study Evaluating Potential Drug-drug Interactions Between Gemfibrozil (Part 1) or Dabigatran Etexilate (Part 2) and Camlipixant (BLU-5937) 50 mg Tablet in Healthy Participants Under Fasting Conditions
Brief Title: Evaluation of the Potential Drug-drug Interactions Between Gemfibrozil or Dabigatran Etexilate and Camlipixant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 221854; BUS-P1-12 (Other: Bellus Health Inc)
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cough; Healthy
MeSH Terms: conditions — Cough | interventions — Dabigatran; Gemfibrozil

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg (Experimental): Participants received a single oral dose of camlipixant 50 milligram (mg) tablet on Day 1, followed by repeat oral doses of gemfibrozil 600 mg tablet twice daily (BID), every 12 hours, (total daily dose of 1200 mg) on Days 5 to 11, with co-administration of a single oral dose of camlipixant 50 mg tablet with the gemfibrozil on Day 9. There was a washout of at least 4 days between the dose of camlipixant on Day 1 and the dose of gemfibrozil on Day 5.
  Interventions: Drug: Camlipixant; Drug: Gemfibrozil
- Part 2: Dabigatran etexilate 150 mg + camlipixant 50 mg (Experimental): Participants received single oral dose of dabigatran etexilate 150 mg capsule on Day 1, followed by repeated oral doses of camlipixant 50 mg tablet twice daily (BID) (total daily dose of 100 mg) from Days 5 to 9, with co-administration of a single oral dose of dabigatran etexilate 150 mg capsule with the morning dose of camlipixant on Day 10. There was a washout of at least 4 days between the dose of dabigatran etexilate on Day 1 and the dose of camlipixant on Day 5.
  Interventions: Drug: Camlipixant; Drug: Dabigatran etexilate

INTERVENTIONS:
Drug: Camlipixant — Camlipixant will be administered
Drug: Dabigatran etexilate — Dabigatran etexilate will be administered
  Arms: Part 2: Dabigatran etexilate 150 mg + camlipixant 50 mg
Drug: Gemfibrozil — Gemfibrozil will be administered.
  Arms: Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg

SUMMARY:
This is a phase 1, 2-part, open-label, fixed-sequence study evaluating potential drug-drug interactions between gemfibrozil (part 1) or dabigatran etexilate (part 2) and camlipixant (BLU-5937) 50 mg tablet in healthy participants under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females

Exclusion Criteria:

* History of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disorder, as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Québec, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 45 participants were enrolled in the study (25 participants in Part 1 and 20 participants in Part 2). Only 32 participants (13 participants were never dosed) were dosed into the study to receive either camlipixant + gemfibrozil or dabigatran etexilate+ camlipixant creating the Safety Population. (The safety population included all participants who received at least one dose of any study drug).
Period: Part 1 (Up to Day 21)
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Started (Enrolled) | 25 | 0
Safety Population | 16 | 0
Completed | 15 | 0
Not Completed | 10 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Enrolled but did not receive study treatment | 9 | 0
Period: Part 2 (Up to Day 22)
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Started (Enrolled) | 0 | 20
Safety Population | 0 | 16
Completed | 0 | 14
Not Completed | 0 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Enrolled but did not receive study treatment | 0 | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the Safety Population which consisted of all participants who received at least one dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Customized [Count of Participants; unit: Participants]
  23 to 54 years | 16 | 16 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 9 | 9 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — "All Other Races" category (Black and Asian where 0<n<11) are combined into one category to maintain participant confidentiality and privacy
  Participants
    All Other Races | 2 | 2 | 4
    White | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC-inf) of Camlipixant
Description: Blood samples were collected at indicated time points for PK analysis of Camlipixant. PK analysis was conducted using standard non-compartmental methods.
Time Frame: Pre-dose, 0.25 , 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15, 18, 24, 48, 72 hours post-dose on Day 1 and Day 9
Population: The PK parameter Population included all participants for whom the Day 1 and Day 9 PK profiles of the camlipixant could be adequately characterized, specifically, when administered alone and in combination with gemfibrozil (Part 1)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Hours*nanograms per milliliter
  Day 1 | 4886.66 (28.69)
  Day 9 | 10642.07 (24.17)

2. Primary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero Until the Last Observed Concentration (AUC[0-t]) of Camlipixant
Description: as for outcome 1
Time Frame: Pre-dose, 0.25 , 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15, 18, 24, 48, 72 hours post-dose on Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Hours*nanograms per milliliter
  Day 1 | 4846.83 (28.84)
  Day 9 | 10541.57 (24.44)

3. Primary Outcome: Part 1: Maximal Observed Concentration (Cmax) of Camlipixant
Description: as for outcome 1
Time Frame: Pre-dose, 0.25 , 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15, 18, 24, 48, 72 hours post-dose on Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Nanograms per milliliter
  Day 1 | 1078 (25.02)
  Day 9 | 1303 (25.65)

4. Primary Outcome: Part 2: AUC(0-Infinity) of Free Dabigatran
Description: Blood samples were collected at indicated time points for PK analysis of Dabigatran. PK analysis was conducted using standard non-compartmental methods.
Time Frame: Pre-dose, 0.25 , 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36, 48, 60, 72 hours post-dose on Day 1 and Day 10
Population: The PK parameter Population included all participants for whom the Day 1 and Day 10 PK profiles of the dabigatran could be adequately characterized, specifically, when administered alone and in combination with camlipixant (Part 2). Only those participants who were measured and analyzed (i.e., contributed data reported in table) were included in 'Overall Number of Participants Analyzed' field.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Hours*nanograms per milliliter
  Day 1 | 943.49 (52.12)
  Day 10 | 1055.20 (43.81)

5. Primary Outcome: Part 2: AUC(0-t) of Free Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Hours*nanograms per milliliter
  Day 1 | 920.18 (53.11)
  Day 10 | 1031.89 (45.03)

6. Primary Outcome: Part 2: Cmax of Free Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Nanograms per milliliter
  Day 1 | 110 (53.53)
  Day 10 | 125 (47.75)

7. Primary Outcome: Part 2: AUC(0-Infinity) of Total Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Hours*nanograms per milliliter
  Day 1 | 1165.82 (52.34)
  Day 10 | 1339.35 (41.21)

8. Primary Outcome: Part 2: AUC(0-t) of Total Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Hours*nanograms per milliliter
  Day 1 | 1139.80 (53.51)
  Day 10 | 1316.80 (41.83)

9. Primary Outcome: Part 2: Cmax of Total Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Nanograms per milliliter
  Day 1 | 135 (54.20)
  Day 10 | 160 (42.42)

10. Secondary Outcome: Part 1: Time to Reach Maximum Observed Concentration (Tmax) of Camlipixant
Description: as for outcome 1
Time Frame: Pre-dose, 0.25 , 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15, 18, 24, 48, 72 hours post-dose on Day 1 and Day 9
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Hours
  Day 1 | 0.750 [0.500 to 2.000]
  Day 9 | 0.750 [0.500 to 2.500]

11. Secondary Outcome: Part 1: Terminal Elimination Half-Life (T1/2) Following Administration of Camlipixant
Description: as for outcome 1
Time Frame: Pre-dose, 0.25 , 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15, 18, 24, 48, 72 hours post-dose on Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Hours
  Day 1 | 5.56 (31.80)
  Day 9 | 9.56 (18.60)

12. Secondary Outcome: Part 1: Percentage of AUC0-Infinity Due to Extrapolation From the Time of the Last Observed Concentration to Infinity (%AUC Extrapolation) of Camlipixant
Description: Blood samples were collected at indicated time points for PK analysis of Camlipixant. PK analysis was conducted using standard non-compartmental methods. Percentage of AUC extrapolation was calculated as [1 - (AUC0-t/AUC0-inf)] * 100.
Time Frame: Pre-dose, 0.25 , 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15, 18, 24, 48, 72 hours post-dose on Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC extrapolation
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Percentage of AUC extrapolation
  Day 1 | 0.58 (104.04)
  Day 9 | 0.59 (109.24)

13. Secondary Outcome: Part 1: Terminal Elimination Rate Constant of Camlipixant (Kel)
Description: as for outcome 1
Time Frame: Pre-dose, 0.25 , 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15, 18, 24, 48, 72 hours post-dose on Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h^-1
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
h^-1
  Day 1 | 0.1247 (31.80)
  Day 9 | 0.0725 (18.60)

14. Secondary Outcome: Part 1: Apparent Clearance (CL/F) of Camlipixant
Description: as for outcome 1
Time Frame: Pre-dose, 0.25 , 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15, 18, 24, 48, 72 hours post-dose on Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Liters per hour
  Day 1 | 10.23 (28.69)
  Day 9 | 4.70 (24.17)

15. Secondary Outcome: Part 1: Apparent Volume of Distribution (Vz/F) of Camlipixant
Description: as for outcome 1
Time Frame: Pre-dose, 0.25 , 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15, 18, 24, 48, 72 hours post-dose on Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Liters
  Day 1 | 82.06 (22.57)
  Day 9 | 64.80 (23.69)

16. Secondary Outcome: Part 2: Tmax of Free Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Hours
  Day 1 | 2.000 [1.500 to 3.500]
  Day 10 | 2.000 [1.500 to 3.000]

17. Secondary Outcome: Part 2: T1/2 Following Administration Free Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Hours
  Day 1 | 10.49 (18.23)
  Day 10 | 9.18 (9.16)

18. Secondary Outcome: Part 2: Percentage of AUC0-Infinity Due to Extrapolation From the Time of the Last Observed Concentration to Infinity (%AUC Extrapolation) of Free Dabigatran
Description: Blood samples were collected at indicated time points for PK analysis of Dabigatran. PK analysis was conducted using standard non-compartmental methods. Percentage of AUC extrapolation was calculated as [1 - (AUC0-t/AUC0-inf)] * 100.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC extrapolation
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Percentage of AUC extrapolation
  Day 1 | 2.22 (49.87)
  Day 10 | 1.95 (52.63)

19. Secondary Outcome: Part 2: Kel Free Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h^-1
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
h^-1
  Day 1 | 0.0660 (18.23)
  Day 10 | 0.0755 (9.16)

20. Secondary Outcome: Part 2: CL/F Free Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Liters per hour
  Day 1 | 158.98 (52.12)
  Day 10 | 142.15 (43.81)

21. Secondary Outcome: Part 2: Vz/F Free Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Liters
  Day 1 | 2407.03 (54.73)
  Day 10 | 1883.56 (43.72)

22. Secondary Outcome: Part 2: Tmax of Total Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Hours
  Day 1 | 2.000 [1.000 to 3.500]
  Day 10 | 2.000 [1.000 to 3.000]

23. Secondary Outcome: Part 2: T1/2 Following Administration of Total Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Hours
  Day 1 | 11.04 (30.01)
  Day 10 | 10.21 (16.90)

24. Secondary Outcome: Part 2: Percentage of AUC0-Infinity Due to Extrapolation From the Time of the Last Observed Concentration to Infinity (%AUC Extrapolation) of Total Dabigatran
Description: as for outcome 18
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC extrapolation
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Percentage of AUC extrapolation
  Day 1 | 1.93 (59.97)
  Day 10 | 1.58 (37.14)

25. Secondary Outcome: Part 2: Kel of Total Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h^-1
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
h^-1
  Day 1 | 0.0628 (30.01)
  Day 10 | 0.0679 (16.90)

26. Secondary Outcome: Part 2: CL/F of Total Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Liters per hour
  Day 1 | 128.66 (52.34)
  Day 10 | 111.99 (41.21)

27. Secondary Outcome: Part 2: Vz/F of Total Dabigatran
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 14
Liters
  Day 1 | 2048.49 (61.16)
  Day 10 | 1649.21 (37.35)

28. Secondary Outcome: Part 1: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs) and Treatment-emergent Adverse Events of Medical Interest (TEAEMIs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant who is administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. Serious adverse events (SAEs) are defined as any untoward medical occurrence that; at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, other situations as per medical and scientific judgement. Adverse events of medical interest (AEMIs) are AEs of scientific interest specific to the drug class. AEMIs for this study includes the following, but not limited to taste disturbances (dysgeusia, hypogeusia, ageusia), oral paresthesia and oral hypoesthesia Treatment-emergent events (i.e., TEAEs, TESAEs and TEAEMIs) were defined as events that commence on or after the time of first study drug administration
Time Frame: Day 1 post-dose until Day 5 pre-dose of gemfibrozil [camlipixant 50mg]; from Day 5 dosing until Day 9 pre-dose of camlipixant [gemfibrozil 600mg]; from camlipixant dosing on Day 9 until end of study [Day 21] [camlipixant 50mg+gemfibrozil 600mg]
Population: Safety Population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Camlipixant 50 mg: Participants received a single oral dose of 50 mg camlipixant tablet on Day 1.
- Part 1: Gemfibrozil 600 mg: Participants received repeated oral doses of gemfibrozil 600 mg tablet twice daily (BID), every 12 hours, (total daily dose of 1200 mg) on Days 5 to 11
- Part 1: Camlipixant 50 mg+ Gemfibrozil 600 mg: Participants received repeated oral doses of gemfibrozil 600 mg tablet twice daily (BID), every 12 hours, (total daily dose of 1200 mg) on Days 5 to 11, with co-administration of a single oral dose of camlipixant 50 mg tablet with the gemfibrozil on Day 9. Participants were followed up for adverse events until end of study (up to Day 21)
Arm/Group | Part 1: Camlipixant 50 mg | Part 1: Gemfibrozil 600 mg | Part 1: Camlipixant 50 mg+ Gemfibrozil 600 mg
Number analyzed (Participants) | 16 | 16 | 16
Participants
  TEAEs | 1 | 6 | 5
  TESAEs | 0 | 0 | 1
  TEAEMIs | 0 | 0 | 1

29. Secondary Outcome: Part 2: Number of Participants With TEAEs, TESAEs and TEAEMIs
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant who is administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. Serious adverse events (SAEs) are defined as any untoward medical occurrence that; at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, other situations as per medical and scientific judgement. Adverse events of medical interest (AEMIs) are AEs of scientific interest specific to the drug class. AEMIs for this study includes the following, but not limited to: taste disturbances (dysgeusia, hypogeusia, ageusia), oral paresthesia and oral hypoesthesia Treatment-emergent events (i.e., TEAEs, TESAEs and TEAEMIs) were defined as events that commence on or after the time of first study drug administration.
Time Frame: Day1 postdose until Day5 predose of camlipixant [dabigatran etexilate 150mg];from Day5 dosing until Day10 predose of dabigatran [camlipixant 50mg];from dabigatran dosing on Day10 until end of study [Day 22][dabigatran etexilate 150mg+camlipixant 50mg]
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Dabigatran Etexilate 150 mg: Participants received single oral dose of dabigatran etexilate 150 mg capsule on Day 1
- Part 2: Camlipixant 50 mg: Participants received repeated oral doses of camlipixant 50 mg tablet twice daily (BID) (total daily dose of 100 mg) from Days 5 to 10
- Part 2: Dabigatran Etexilate 150 mg+ Camlipixant 50 mg: Participants received repeated oral doses of camlipixant 50 mg tablet twice daily (BID) (total daily dose of 100 mg) from Days 5 to 9, with co-administration of a single oral dose of dabigatran etexilate 150 mg capsule with the morning dose of camlipixant on Day 10. Participants were followed up for adverse events until end of study (up to Day 22)
Arm/Group | Part 2: Dabigatran Etexilate 150 mg | Part 2: Camlipixant 50 mg | Part 2: Dabigatran Etexilate 150 mg+ Camlipixant 50 mg
Number analyzed (Participants) | 16 | 15 | 14
Participants
  TEAEs | 4 | 6 | 0
  TESAEs | 0 | 0 | 0
  TEAEMIs | 0 | 0 | 0

30. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in 12-Lead Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was recorded with the participant in a semi-recumbent or supine position, after 5 minutes of rest using an ECG machine. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for the number of participants with abnormal clinically significant 12-Lead ECG findings have been presented.
Time Frame: Day 5, Day 9 pre-dose and 1 hour post-dose, Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Participants
  Day 5 | 0
  Day 9, Pre-dose | 0
  Day 9,1-Hour Post-dose | 0
  Day 12 | 0

31. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in 12-Lead ECG Findings
Description: as for outcome 30
Time Frame: Day 5, Day 10 and Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 16
Participants
  Day 5 | 0
  Day 10 | 0
  Day 13 | 0

32. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Vital Signs: Diastolic Blood Pressure (DBP), Systolic Blood Pressure (SBP), and Heart Rate
Description: Vital signs including DBP, SBP, and heart rate were measured in a sitting position after resting for at least 5 minutes. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for the number of participants with abnormal clinically significant changes for vital signs have been presented.
Time Frame: Day 9 and Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Participants
  Day 9 | 0
  Day 12 | 0

33. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Vital Signs: DBP, SBP, and Heart Rate
Description: as for outcome 32
Time Frame: Day 10 and Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 16
Participants
  Day 10 | 0
  Day 13 | 0

34. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Vital Signs: Respiratory Rate and Oral Temperature
Description: Vital signs including respiratory rate and oral temperature were measured after resting for at least 5 minutes in a sitting position. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for the number of participants with abnormal clinically significant changes for vital signs have been presented.
Time Frame: Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Participants | 0

35. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Vital Signs: Respiratory Rate and Oral Temperature
Description: as for outcome 34
Time Frame: Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 16
Participants | 0

36. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes During Physical Examination
Description: Physical examination included assessment of the head, eyes, ears, nose, throat, neck, chest, lungs, abdomen, musculoskeletal, dermatological, cardiovascular/peripheral vascular, and general neurological examination. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for the number of participants with abnormal clinically significant changes in physical examination has been presented.
Time Frame: Up to Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Participants | 1

37. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes During Physical Examination
Description: as for outcome 36
Time Frame: Up to Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 16
Participants | 0

38. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Hematology Parameters
Description: Blood samples were collected to analyze hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Hematocrit, Hemoglobin, Platelets, and Erythrocytes. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Number of participants with abnormal clinically significant changes in hematology parameters were reported.
Time Frame: Up to Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Participants | 0

39. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Hematology Parameters
Description: as for outcome 38
Time Frame: Up to Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 16
Participants | 0

40. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Clinical Chemistry Parameters
Description: Blood samples were collected to analyze clinical chemical parameters: albumin, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, calcium, chloride, creatinine kinase, creatinine, gamma glutamyl transferase, glucose, phosphate, potassium, sodium, total, direct, and indirect bilirubin, protein, urea, and urate. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Number of Participants with abnormal clinically significant changes in clinical chemistry parameters were reported.
Time Frame: Up to Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Participants | 3

41. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Clinical Chemistry Parameters
Description: as for outcome 40
Time Frame: Up to Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 16
Participants | 1

42. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Coagulation Parameters
Description: Blood samples were collected to analyze coagulation parameters: activated partial thromboplastin time, prothrombin time international normalized ratio (INR), and prothrombin time. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Number of Participants with abnormal clinically significant changes in coagulation parameters were reported.
Time Frame: Up to Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Participants | 0

43. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Coagulation Parameters
Description: as for outcome 42
Time Frame: Up to Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 16
Participants | 0

44. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Urinalysis
Description: Urine samples were collected to analyze urinalysis parameters: specific gravity and potential of hydrogen (pH). Bilirubin, blood (occult), glucose, ketones, leukocyte esterase, nitrite, protein, urobilinogen were analyzed by dipstick. The dipstick test gives results in a semi-quantitative manner, and results can be read as Negative, Trace, 1+, 2+ indicating proportional concentrations in the urine sample. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Number of Participants with abnormal clinically significant changes in urinalysis parameters were reported.
Time Frame: Up to Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Gemfibrozil 600 mg
Number analyzed (Participants) | 16
Participants | 0

45. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Urinalysis
Description: as for outcome 44
Time Frame: Up to Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Dabigatran Etexilate 150 mg + Camlipixant 50 mg
Number analyzed (Participants) | 16
Participants | 0

ADVERSE EVENTS:
Time Frame: Part1(Day1 postdose until Day5 predose of gemfibrozil [Camlipixant 50mg];from Day5 dosing until Day9 predose of camlipixant[Gemfibrozil 600mg];from camlipixant dosing on Day9 until end of study[Day21] [Camlipixant 50mg+Gemfibrozil 600mg]) and Part2(Day1 postdose until Day5 predose of camlipixant[Dabigatran etexilate 150mg];from Day5 dosing until Day10 predose of dabigatran[Camlipixant 50mg];from dabigatran dosing on Day10 until end of study [Day22] [Dabigatran etexilate 150mg+camlipixant 50mg])
Description: Safety Population comprised of all participants who received at least one dose of any study drug. AEs were reported treatment-wise.
Arm/Group | Part 1: Camlipixant 50 mg | Part 1: Gemfibrozil 600 mg | Part 1: Camlipixant 50 mg+ Gemfibrozil 600 mg | Part 2: Dabigatran Etexilate 150 mg | Part 2: Camlipixant 50 mg | Part 2: Dabigatran Etexilate 150 mg+ Camlipixant 50 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 1/16 | 0/16 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 1/16 | 6/16 | 5/16 | 4/16 | 6/15 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Camlipixant 50 mg (N=16) | Part 1: Gemfibrozil 600 mg (N=16) | Part 1: Camlipixant 50 mg+ Gemfibrozil 600 mg (N=16) | Part 2: Dabigatran Etexilate 150 mg (N=16) | Part 2: Camlipixant 50 mg (N=15) | Part 2: Dabigatran Etexilate 150 mg+ Camlipixant 50 mg (N=14)
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Camlipixant 50 mg (N=16) | Part 1: Gemfibrozil 600 mg (N=16) | Part 1: Camlipixant 50 mg+ Gemfibrozil 600 mg (N=16) | Part 2: Dabigatran Etexilate 150 mg (N=16) | Part 2: Camlipixant 50 mg (N=15) | Part 2: Dabigatran Etexilate 150 mg+ Camlipixant 50 mg (N=14)
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thyroxine free decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT05959447/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT05959447/SAP_001.pdf